CLINICAL TRIAL: NCT04503239
Title: Prediabetes and Type 2 Diabetes Data Collection Study: T2Help
Brief Title: Prediabetes and Type 2 Diabetes Data Collection Study
Acronym: T2Help
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-904050
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus, Type 2; Pre-diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (9):
- Prediabetes (both IGT and IFG): Device: G6 Participant to wear G6 and activity tracker for 3 months and add meals and medications into e-diary daily
  Interventions: Device: G6
- Type 2 Diabetes on 1 OAD: Participant to wear G6 and activity tracker for 3 months and add meals and medications into e-diary daily
  Interventions: Device: G6
- Type 2 Diabetes on 2 or more OAD: Participant to wear G6 and activity tracker for 3 months and add meals and medications into e-diary daily
  Interventions: Device: G6
- Type 2 Diabetes using Basal insulin with or without OAD: Participant to wear G6 and activity tracker for 3 months and add meals and medications into e-diary daily
  Interventions: Device: G6
- Type 2 Diabetes in GLP-1 with or without OAD: Participant to wear G6 and activity tracker for 3 months and add meals and medications into e-diary daily
  Interventions: Device: G6
- Type 2 Diabetes using intense insulin treatment-Multiple Dail: Participant to wear G6 and activity tracker for 3 months and add meals and medications into e-diary daily
  Interventions: Device: G6
- Type 2 Diabetes in MDI or basal insulin plus GLP-1: Participant to wear G6 and activity tracker for 3 months and add meals and medications into e-diary daily
  Interventions: Device: G6
- Type 2 Diabetes on 0 OAD: Participant to wear G6 and activity tracker for 3 months and add meals and medications into e-diary daily
  Interventions: Device: G6
- High Risk to Develop Prediabetes / Type 2 Diabetes: Participant to wear G6 and activity tracker for 3 months and add meals and medications into e-diary daily
  Interventions: Device: G6

INTERVENTIONS:
Device: G6 — Wear 9 wear periods of the 10-day CGM

SUMMARY:
To collect data in an observational study from Prediabetes (PD) and Type 2 Diabetes (T2D) patients including time correlated CGM, medication and food intake approximately 80% of the time for each subject that completes the entire active phase.

DETAILED DESCRIPTION:
In addition, lifestyle and treatment already established for prediabetes and Type 2 Diabetes such as:

* Sleep
* Exercise/Physical activity/or lack of it
* Heart rate
* Five hours OGTT- 6 subjects in each group that have C-Peptide positive lab result at screening and consent to the OGTT (Appendix 3) This data will address the sources and nature of blood glucose variability across the progression of PD and T2D. The data collected in this study will enable investigation into CGM-data artifacts that speak to the state and management of PD and T2D. Possible applications enabled by these data sets include: compliance with drug regimens and other lifestyle recommendations, drug titration and/or escalation/de-escalation, and diagnosis and/or treatment throughout the progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ages ≥18 years of age at the time of screening
* High Risk of developing PD or T2D with HbA1c ≤5.6%

With one or more of the following:

* Strong family history of T2D
* BMI ≥35 kg/m2
* History of gestational diabetes mellitus (GDM)
* Age and Race, Ethnicity
* Polycistic Ovarian Syndrome
* High Blood Pressure
* Abnormal cholesterol and triglyceride levels

  * Clinical Diagnosis of Prediabetes (PD) as defined by ADA to have an HbA1c ≥5.7%-6.4%. or clinical diagnosis of Type 2 Diabetes (T2D) with HbA1c between ≥6.5 % and ≤12.0%. Determined via medical record or source documentation by an individual qualified to make a medical diagnosis.
  * Having no treatment, one or more of the combination of treatments for the disease in every spectrum such as exercise and diet for PD and no treatment, 1 or more methods of treatment for T2D and combination of treatments for the disease MDI or CSII alone, MDI or CSII plus OAD and MDI or CSII with or without GLP-1 with or without OAD.
  * No change in diabetic medication in the last three months for patients in treatment.
  * Willingness to use a study provided CGM, use of an activity tracker, and agree to record data related to food and medication intake in an e-diary (e.g. mobile app).
  * For a subset of subjects who agree to provide consent, an OGTT will be performed as explained on Appendix 3. OGTT will be performed on 6 subjects per group that have a lab result with positive c-peptide. Having a smartphone compatible with Dexcom G6 CGM, activity tracker & e-Diary. (This could be provided by the study team if the qualified subject does not have smartphone compatible with apps. For users that do not use their personal smartphones for data collection purposes, the T2Help study will provide a commercially available smartphone. The smartphones will be modified so they are only capable of hosting and running the study applications required for data collection (Fitbit, Welldoc, G6). The modified smartphones will not be able to execute standard smartphone functionality such as internet browsing, texting, or making phone calls. Bluetooth functionality will remain intact as it is required for the approved applications to collect data.)
  * If using additional medication, such as thyroid, hypertension, and cholesterol lowering medication these have to be stable for at least 3 months.

Exclusion Criteria:

* Hospital admissions for diabetes ketoacidosis (DKA) or Hyperglycemic Hyperosmolar Nonketotic Syndrome (HHNS) in the last 6 months.
* History of 2 or more episodes of severe hypoglycemia, which resulted in any of the following during the 6 months prior to screening:

Medical assistance by a third party (Caregiver needed to inject glucagon, ER visit, hospitalization) Coma Seizures

* Subject has a skin condition for which he/she is unable to tolerate tape adhesive in the area of sensor placement.
* Pregnancy (as demonstrated by a positive test at study entry) at time of screening or are planning to become pregnant during the study.
* Subject has had any of the following cardiovascular events within 3 months of screening: myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, recent transient ischemic attack, cerebrovascular accident with sequelae, unstable angina, unstable congestive heart failure, unstable ventricular rhythm disturbances or thromboembolic disease.
* Unstable thyroid disease. (changes in Thyroid medication in the last 90 days)
* Subject has taken any oral, injectable, or intravenous (IV) steroids within 8 weeks from the time of screening visit, or plans to take any oral, injectable, or IV steroids during the course of the study.
* Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks.
* Subject is currently using illicit drugs.
* Subject is currently abusing prescription drugs.
* Subject is currently abusing alcohol.
* Subject has a history of visual impairment which would not allow him/her to participate in the study and perform all study procedures safely, as determined by the investigator.
* Subject has elective surgery planned that requires general anesthesia during the course of the study.
* Subject has a sickle cell disease, hemoglobinopathy, or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening.
* Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation.
* Subject diagnosed with current eating disorder such as anorexia or bulimia.
* Subject is on dialysis.
* Subject has eGFR <45 confirmed by medical record.
* Recent Pancreatitis. (< 30 days)
* Cancer/malignancy in treatment.
* Cystic fibrosis.
* Any other problem for which the investigator or the sponsor may believe that the subject will not be able to comply with the study. (e.g. use of hydroxyurea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — not pregnant or planning on becoming pregnant during study
Study Population: Pre-diabetics and Type 2 Diabetics 18 and over willing to wear 2 study devices and enter in the daily medication and food intake.
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-02-27 (Estimated); Study Completion 2022-02-27 (Estimated)

PRIMARY OUTCOMES:
Collect Device Data - CGM | up to 16 weeks
  To collect data in an observational study from Prediabetes (PD) and Type 2 Diabetes (T2D) patients including time correlated CGM approximately 80% of the time for each subject that completes the entire active phase.
Collect Device Data - e-Diary | up to 16 weeks
  To collect data in an observational study from Prediabetes (PD) and Type 2 Diabetes (T2D) patients including logging diabetic medication taken or not taken 80% of the time for each subject that completes the entire active phase.
Collect Device Data - e-Diary | up to 16 weeks
  To collect data in an observational study from Prediabetes (PD) and Type 2 Diabetes (T2D) patients including logging food intake approximately 80% of the time for each subject that completes the entire active phase.
Collect Device Data - Activity Tracker | up to 16 weeks
  To collect data in an observational study from Prediabetes (PD) and Type 2 Diabetes (T2D) patients including logging lifestyle by activity tracker approximately 80% of the time for each subject that completes the entire active phase.

SECONDARY OUTCOMES:
Collect Current Subject Lifestyle and Treatment Regimen | up to 16 weeks
  Collect subjects current treatment already established for Prediabetes and Type 2 Diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Danny Chernavvsky, MD, Study Director — DexCom, Inc.
Locations (5):
- United States (5):
  - Synergy San Diego, Lemon Grove, California
  - Palm Research Center, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Diabetes and Glandular Disease, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No